CLINICAL TRIAL: NCT04016610
Title: Proof of Concept (POC) Study of the Soliton's Acoustic Scar Reduction (ASR) Treatment Using Rapid Acoustic Pulse (RAP) Device for the Treatment of Keloid Scar
Brief Title: Proof of Concept (POC) Study of the Soliton's Acoustic Scar Reduction (ASR) Treatment for the Treatment of Keloid Scar
Acronym: ASR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Collaborators: Emergent Clinical Consulting, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Soliton 2019-001
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Keloid Scar
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ASR Treatment (Experimental): Single and/or multi-treatment ASR device applied to the keloid scar for a period of 2 minutes for each 3 cm.
  Interventions: Device: Soliton's Acoustic Scar Reduction (SAR)

INTERVENTIONS:
Device: Soliton's Acoustic Scar Reduction (SAR) — Treatment of keloid scars for the temporary improvement in appearance.

SUMMARY:
To evaluate the safety, and efficacy of the ASR device for the temporary improvement in the appearance of a keloids.

DETAILED DESCRIPTION:
To evaluate the safety, and efficacy of the ASR device for the temporary improvement in the appearance of a keloids. To demonstrate improvement in the keloid scars, without unexpected adverse events (UAEs) and serious adverse events (SAEs) directly attributable to the ASR device or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 18 at the screening visit;
* The participant is healthy, as determined by the investigator based on a medical evaluation including medical history;
* The participant has a keloid that is easily delineated photographically located on the chest, back, trunk or upper arms and legs.
* Keloid size greater than 1 cm and less than 8 cm in length, with a height of at least 2 mm.
* Keloids less than 5 years old
* Body Mass Index (B.M.I.) is > 20
* Participant is willing to not undergo any other keloid treatments for a period of 12 months following ASR treatment.
* Participant is willing to participate in study and adhere to follow-up schedule.
* Participant is able to read and comprehend English or Spanish.
* Participant has completed the Informed Consent Form.

Exclusion Criteria:

* Participant had treatments, including topical steroids, to the keloid being treated in the study in the prior 12 months.
* Participant is unwilling to have research photos taken of treatment areas in the presence of Sponsor's researchers.
* Participant is unwilling to have ASR treatment provided in the presence of Sponsor's researchers.
* Participant is pregnant or planning to become pregnant during the duration of the study.
* Metal or plastic implants near the area of the treatment (vascular stent, plates and screws, chest wires, hips, elbows, knees, etc.).
* Active electronic implants such as pacemakers, defibrillators, cochlear implants, nerve/brain stimulators, drug pump, etc.
* Medical disorder that would hinder the wound healing or immune response (no blood disorder, etc.).
* History of coagulopathy(ies) and/or on anticoagulant medication.
* Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
* Current smoker.
* Any surgical procedure in the prior 3 months, or planned during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Procedure Safety | 12 weeks
  The safety endpoint will be met if all treated participants are free from unexpected adverse events and serious adverse events directly attributable to the ASR device or treatment.

SECONDARY OUTCOMES:
Treatement Tolerability | 12 weeks
  ASR treatment tolerability will be met if the average pain measure using a 0-10 pain scale across all treated Participants is < 8.0.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Capelli, MD, Study Director — Soliton, Inc.
Locations (1):
- Clear Dermatology and Aesthetics Center, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No